CLINICAL TRIAL: NCT00419263
Title: A Phase II, Multicenter, Randomized, Double-Mask, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Intramuscular Peramivir in Subjects With Uncomplicated Acute Influenza.
Brief Title: Evaluation of the Efficacy and Safety of Peramivir in Subjects With Uncomplicated Acute Influenza.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCX1812-211
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-01

CONDITIONS: Influenza
Keywords: influenza; flu
MeSH Terms: conditions — Influenza, Human | interventions — peramivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Peramivir 150 mg (Experimental)
  Interventions: Drug: Peramivir 150 mg
- Peramivir 300 mg (Experimental)
  Interventions: Drug: Peramivir 300 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Peramivir 150 mg — Single dose administered as bilateral 2-mL intramuscular injections in each gluteal muscle (one injection of peramivir 150 mg and one injection of placebo).
  Other Names: BCX1812
  Arms: Peramivir 150 mg
Drug: Peramivir 300 mg — Single dose administered as bilateral 2-mL intramuscular injections in each gluteal muscle (2 injections of peramivir 150 mg).
  Other Names: BCX1812
  Arms: Peramivir 300 mg
Drug: Placebo — Single dose administered as bilateral 2-mL intramuscular injections in each gluteal muscle (2 injections of placebo).
  Arms: Placebo

SUMMARY:
This is a study for patients with flu who also have a fever as well as other flu symptoms. Patients must have had symptoms for less than 48 hours in order to participate. Patients will have two out of three chances of getting an active study treatment and the other third will receive a placebo (dummy drug). Nobody will know who gets the active drug and who gets the inactive drug. All patients will get supplies to treat symptoms of flu. Patients will need to be seen 5 more times after they are enrolled in the study.

DETAILED DESCRIPTION:
Peramivir is a neuraminidase inhibitor that was previously shown to be effective in the treatment of human experimental influenza using an oral formulation. Parenteral formulations of peramivir (for intramuscular and intravenous injection) entered clinical development at the time of this Phase 2 study. A series of Phase 1 studies in human volunteers was completed that provided safety and pharmacokinetic results that supported the initiation of this Phase 2 multinational, randomized, double-mask study that compared the antiviral efficacy and safety of peramivir administered intramuscularly versus placebo in adults with uncomplicated acute influenza. Because of the unique pharmacokinetic and pharmacodynamic properties of peramivir - a long terminal half life in plasma and an extended duration of binding to the neuraminidase enzyme - subjects were randomized in a 1:1:1 ratio to receive a single dose of one of three treatments: peramivir 150 mg, peramivir 300 mg, and placebo. Study drug was administered as one 2-mL intramuscular injection in each gluteal muscle (total of 4 mL, injected in divided doses). This multinational study was originally to be conducted at approximately 80 sites in the US and Canada. When enrollment during the North American influenza season of 2006-2007 did not achieve the target, the study was extended to sites in Australia, New Zealand, South Africa, and Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Presence of fever at time of screening of ≥38.0 ºC (≥100.4 ºF) taken orally, or ≥38.5 ºC (≥101.2 ºF) taken rectally. However, this requirement is waived if the subject has a history of fever within the 24 hours prior to screening and has been administered antipyretic(s) in the 6 hours prior to screening.
* Presence of at least one respiratory symptom (cough, sore throat, or nasal symptoms) of any severity (mild, moderate, or severe)
* Presence of at least one constitutional symptom (headache, malaise, myalgia, sweats and/or chills, or fatigue) of any severity (mild, moderate, or severe)
* Onset of illness no more than 48 hours before presentation. Note: Time of onset of illness is defined as either (1) the time when the temperature (either oral or rectal) was first measured as elevated (at least one ºC of elevation-oral temperature), OR (2) the time when the subject experienced the presence of at least one respiratory symptom AND the presence of at least one constitutional symptom.
* Rapid Antigen Test (RAT) performed on an adequate specimen collected from an anterior nasal swab is positive. A negative initial RAT may be repeated within one hour of obtaining a negative result. A second negative RAT result will exclude the subject from evaluation for enrollment.
* Females of childbearing potential must report one of the following:

  * Be surgically sterile
  * Have been sexually abstinent 4 weeks prior to date of screening evaluation and be willing to remain abstinent through 4 weeks after study drug administration
  * Use oral contraceptives or other form of hormonal birth control including hormonal vaginal rings or transdermal patches and have been using these for 3 months prior through 4 weeks after study drug administration
  * Use an intra-uterine device (IUD), or adequate barrier contraception (or double-barrier method such as condom or diaphragm with spermicidal gel or foam) as birth control 4 weeks prior to date of screening evaluation through 4 weeks after study drug administration.

Exclusion Criteria:

* Women who are breast-feeding
* History of diagnosed chronic obstructive pulmonary disease or diagnosis of severe persistent asthma
* History of chronic renal impairment requiring hemodialysis or known or suspected to have moderate or severe renal impairment (actual or estimated creatinine clearance <50 mL/min)
* History of congestive heart failure requiring daily pharmacotherapy with symptoms consistent with New York Heart Association Class II, III, or IV within the past 12 months
* Immunocompromised status due to illness or previous organ transplant
* Current use of systemic immunosuppressive medications (except inhaled corticosteroids)
* Use of rimantadine, amantadine, zanamivir, or oseltamivir in the past 7 days
* Immunized against influenza with live attenuated virus vaccine (FluMist®) in the previous 21 days
* Clinical evidence of active bacterial infection at any body site requiring therapy with oral or systemic antibiotics
* Clinically significant signs of acute respiratory distress
* Clinically significant signs of acute cardiac disease
* Screening ECG which suggests acute ischemia or presence of medically significant dysrhythmia
* Presence of a chronic disease or illness(es) with either clinical or historical evidence of recent exacerbation of such disease(s) or illness(es) or lack of control of such disease(s) or illness(es)
* History of hepatitis B, hepatitis C, or human immunodeficiency virus infection
* History of alcohol abuse or drug addiction within 1 year prior to admission in the study
* Participation in a study of any investigational drug within the last 30 days
* Positive urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Block, MD, Principal Investigator — Kentucky Pediatric/Adult Research; James Borders, MD, Principal Investigator — Central Kentucky Research Assoc, Inc; Robert Broker, MD, Principal Investigator — Hillcrest Family Practice; Paul Browstone, MD, Principal Investigator — Alpine Clinical Research Center; Jeffry Jacqmein, MD, Principal Investigator — Jacksonville Center For Clinical Research; Isaac Marcadis, MD, Principal Investigator — Palm Beach Research Center; Mark Stich, MD, Principal Investigator — Jacksonville Center For Clinical Research; George Atiee, MD, Principal Investigator — GSA Research; Joe Blumenau, MD, Principal Investigator — Research Across America; John Champlin, MD, Principal Investigator — Medical Center; Shane Christensen, MD, Principal Investigator — J. Lewis Research, Inc. Foothill Family Clinic South; Steven Duckor, MD, Principal Investigator — Advanced Clinical Research Institute; Lewis Eirinberg, MD, Principal Investigator — Midwest Family Physicians; Milton K. Erman, MD, Principal Investigator — Pacific Sleep Medicine Services; Stanley Cohen, MD, Principal Investigator — Radiant Research; David L. Fried, MD, Principal Investigator — Omega Medical Research; Yury Furman, MD, Principal Investigator — Pacific Sleep Medicine Services, Inc.; Wayne Harper, MD, Principal Investigator — Wake Research Associates, LLC; Dan C Henry, MD, Principal Investigator — J. Lewis Research, Inc. Foothill Family Clinic; John M. Hill, MD, Principal Investigator — University Clinical Research-Deland, LLC; Veryl Hodges, DO, Principal Investigator — Clopton Clinic; Reuben Holland, III, MD, Principal Investigator — Clinical Research Center; William Jennings, MD, Principal Investigator — Radiant Research San Antonio; James Edmond Kelaher, MD,MPH, Principal Investigator — Baylor Clinic-Baylor College of Medicine; Allan Kelly, MD, Principal Investigator — Hermitage Medicentres; Ben Lasko, MD, Principal Investigator — Manna Research; Mark Leber, MD, Principal Investigator — The Brooklyn Hospital Center; Larissa Lim, MD, Principal Investigator — Florida Medical Research Institute; Alain Martel, MD, Principal Investigator — Clinique medicale des Campus; Dennis Mikolich, MD, Principal Investigator — Paragon Clinical Research, Inc.; Julie Mullen, MD, Principal Investigator — Sterling Research Group, LTD.; David Parenti, MD, Principal Investigator — George Washington University; Monica Pierson, MD, Principal Investigator — Radiant Research; Robert Poirier, MD, Principal Investigator — Barnes-Jewish Hospital Emergency Department; Ivan Rarick, MD, Principal Investigator — Benchmark Research; Dennis Riff, MD, Principal Investigator — Advanced Clinical Research Institute; Q Rizvi, MD, Principal Investigator — Castledowns Medicentre; Michael Rokeach, MD, Principal Investigator — Pacific Sleep Medicine Services; Rawle Seupaul, MD, Principal Investigator — Wishard Hospital; Daniel Shu, MD, Principal Investigator — Gain Medical Research Centre; Steve Sitar, MD, Principal Investigator — Orange County Clinical Trials; Kirk Stiffler, MD, Principal Investigator — Summa Emergency Associates Inc.; Guy Tellier, MD, Principal Investigator — Omnispec clinical research Inc; Michael Warren, MD, Principal Investigator — Research Across America at Oyster Point Family Health Center; Randall Watson, MD, Principal Investigator — J. Lewis Research, Inc./Southwest Family Medicine; John Michael Wise, MD, Principal Investigator — Bozeman Urgent Care Center; Chivers Woodruff, Jr., MD, Principal Investigator — Radiant Research; Bruce Berwald, MD, Principal Investigator — Radiant Research; Frank Maggiacomo, DO, Principal Investigator — New England Center for Clinical Research, Inc; Barry Packman, MD, Principal Investigator — Radiant Research; Sheila Rodstein, MD, Principal Investigator — Radiant Research, Minneapolis; Bernardo Ng, MD, Principal Investigator — Pacific Sleep Medicines Service; Gerardo Losoya, MD, Principal Investigator — Towngate Plaza Medical Center; Francis X. Burch, MD, Principal Investigator — Radiant Research-San Antonio Northeast; John P. Delgado, MD, Principal Investigator — Integrated Medical Research, PC; Edward Fein, MD, Principal Investigator — Pulmonary & Critical Care Associates; Bruce D. Forney, MD, Principal Investigator — Alliance Medical Center; James E. Greenwald, MD, Principal Investigator — Medex Healthcare Research, Inc.; Robert Hudrick, DO, Principal Investigator — University of Medicine & Dentistry of New Jersey; Robert Jeanfreau, MD, Principal Investigator — Benchmark Research; Robert Kaufmann, MD, Principal Investigator — Georgia Clinical Research; Sy Lam, MD, Principal Investigator — Calgary West Medical Centre Clinical Studies; Keith S. Reisinger, MD, MPH, Principal Investigator — Primary Physicians Research, Inc; Keith S. Reisinger, MD, MPH, Principal Investigator — Family Practice Medical Associates South; Earl Martin, MD, Principal Investigator — Dynamed Clinical Research; Jean-Sebastien Gauthier, MD, Principal Investigator — Q & T Research Inc.; Jeffrey Rosen, MD, Principal Investigator — Clinical Research of Southern Florida; Gerald Burns, MD, Principal Investigator — New Orleans Medical; Stewart Behiel, MD, Principal Investigator — Belvedere Medicentre; Giuseppe D'Ignazio, MD, Principal Investigator — Source Unique Clinic; Indravadan Dattani, MD, Principal Investigator — Prairie Clinical; Roy A. Gritter, MD, Principal Investigator — RJA Medicentres; Balbir Chahal, MD, Principal Investigator — Balbir Chahal M.D. ,P.A.
Locations (68):
- United States (57):
  - Radiant Research, Birmingham, Alabama
  - Clopton Clinic, Jonesboro, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Orange County Clinical Trials, Anaheim, California
  - Medical Center, Carmichael, California
  - Pacific Sleep Medicines Service, El Centro, California
  - Advanced Clinical Research Institute, Orange, California
  - Benchmark Research, Sacramento, California
  - Pacific Sleep Medicine Services, San Diego, California
  - Pacific Sleep Medicine Services, San Francisco, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - George Washington Unviersity, Washington D.C., District of Columbia
  - Clinical Research of Southern Florida, Coral Gables, Florida
  - University Clinical Research-Deland, LLC, DeLand, Florida
  - Florida Medical Research Institute, Gainesville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Research Center, Sarasota, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Georgia Clinical Research, Atlanta, Georgia
  - Wishard Hospital, Indianapolis, Indiana
  - Radiant Research, Overland Park, Kansas
  - Kentucky Pediatric / Adult Research, Bardstown, Kentucky
  - Central Kentucky Research Assoc, Inc, Lexington, Kentucky
  - Benchmark Research, Metairie, Louisiana
  - Radiant Research, Minneapolis, Edina, Minnesota
  - Barnes-Jewish Hospital Emergency Department, St Louis, Missouri
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Radiant Research, St Louis, Missouri
  - Bozeman Urgent Care Center, Bozeman, Montana
  - Alliance Medical Center, Alliance, Nebraska
  - Midwest Family Physicians, Omaha, Nebraska
  - UMDNJ, Cherry Hill, New Jersey
  - Pulmonary & Critical Care Associates, East Brunswick, New Jersey
  - Brooklyn Hospital Center, Brooklyn, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Summa Health, Akron, Ohio
  - Sterling Research Group, LTD., Cincinnati, Ohio
  - Integrated Medical Research, PC, Ashland, Oregon
  - Research Across America at Oyster Point Family Health Center, Lancaster, Pennsylvania
  - Radiant Research, Philadelphia, Pennsylvania
  - Primary Physicians Research, Inc, Pittsburgh, Pennsylvania
  - New England Center for Clinical Research, Inc, Cranston, Rhode Island
  - Paragon Clinical Research, Inc., Cranston, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Hillcrest Family Practice, Simpsonville, South Carolina
  - Research Across America, Dallas, Texas
  - Radiant Research, Dallas, Texas
  - Towngate Plaza Medical Center, Garland, Texas
  - Baylor Clinic-Baylor College of Medicine, Houston, Texas
  - GSA Research, San Antonio, Texas
  - Radiant Research-San Antonio Northeast, San Antonio, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - Balbir Chahal M.D. ,P.A, Tomball, Texas
  - Dynamed Clinical Research, Tomball, Texas
  - J. Lewis Research, Inc. Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc./Southwest Family Medicine, West Jordan, Utah
- Canada (11):
  - Calgary West Medical Cnetre Clinical Studies, Calgary, Alberta
  - Belvedere Medicentre, Edmonton, Alberta
  - Hermitage Medicentres, Edmonton, Alberta
  - RJA Medicentres, Edmonton, Alberta
  - Castledowns Medicentre, Edmonton, Alberta
  - Gain Medical Centre, Coquitlam, British Columbia
  - Source Unique Clinic, Hawkesbury, Ontario
  - Manna Research, Toronto, Ontario
  - Omnispec Clinical Reasearch Inc, Mirabel, Quebec
  - Clinique Medicale des Campus, Ste-Foy, Quebec
  - Prairie Clinical, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Peramivir 150 mg | Peramivir 300 mg
Started | 115 | 114 | 115
Completed | 112 | 112 | 112
Not Completed | 3 | 2 | 3
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Randomized in Error, Not Treated | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all subjects who received any dose of study drug. Subjects were analyzed according to the treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Peramivir 150 mg | Peramivir 300 mg | Total
Number analyzed (Participants) | 114 | 113 | 115 | 342
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (12.05) | 36.2 (15.59) | 36.2 (13.25) | 35.4 (13.71)
Age, Customized [Number; unit: participants]
  18 - 27 years old | 41 | 37 | 34 | 112
  28 - 37 years old | 37 | 31 | 35 | 103
  38 - 47 years old | 19 | 21 | 25 | 65
  48 - 57 years old | 9 | 10 | 12 | 31
  ≥ 58 years old | 8 | 13 | 9 | 30
  Missing | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 67 | 62 | 183
  Male | 60 | 46 | 53 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 4 | 19
  Not Hispanic or Latino | 108 | 104 | 111 | 323
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 4 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 6 | 8 | 4 | 18
  Black or African American | 21 | 18 | 17 | 56
  White | 77 | 78 | 81 | 236
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 6 | 14
Body Mass Index at Screening [Mean (Standard Deviation); unit: kg/m^2] — Data were available for 114 participants in the placebo arm, 113 participants in the peramivir 150-mg arm, and 115 participants in the peramivir 300-mg arm.
  kg/m^2 | 26.5 (5.69) | 27.5 (6.23) | 27.8 (6.35) | 27.2 (6.11)
Current Smoking Behavior at Randomization [Number; unit: participants]
  Smoker | 26 | 22 | 25 | 73
  Nonsmoker | 88 | 91 | 90 | 269
Estimated Time of Onset of Symptoms at Screening [Number; unit: participants]
  0 - 12 hours ago | 1 | 4 | 4 | 9
  > 12 - 24 hours ago | 37 | 32 | 25 | 94
  > 24 - 36 hours ago | 45 | 43 | 46 | 134
  > 36 - 48 hours ago | 31 | 34 | 40 | 105
Initial Composite Symptom Score [Mean (Standard Deviation); unit: units on a scale] — Initial Composite Symptom Score is defined as the sum of the 7 symptoms of influenza initially recorded by the subject in the diary (cough; sore throat; nasal congestion; myalgia [aches and pains]; headache; feverishness; and fatigue), each graded on a 4-point severity scale [0, absent; 1, mild; 2, moderate; 3, severe]); for the composite score, individual scores were summed, with a range from 0 to 21. Data were available for 111 participants in the placebo arm, 111 participants in the peramivir 150-mg arm, and 114 participants in the peramivir 300-mg arm.
  units on a scale | 14.3 (3.70) | 14.3 (3.22) | 14.1 (3.92) | 14.2 (3.62)
Influenza Infection [Number; unit: participants] — Infection as measured by polymerase chain reaction (PCR) or serology.
  participants
    Negative | 5 | 9 | 9 | 23
    Positive | 109 | 104 | 105 | 318
    Missing | 0 | 0 | 1 | 1
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Data were available for 114 participants in the placebo arm, 113 participants in the peramivir 150-mg arm, and 115 participants in the peramivir 300-mg arm.
  m^2 | 1.9 (0.26) | 1.9 (0.25) | 1.9 (0.28) | 1.9 (0.26)

OUTCOME MEASURES:

1. Primary Outcome: Time to Alleviation of Symptoms (Kaplan-Meier Estimate)
Description: Descriptive statistics for the primary efficacy variables were tabulated by treatment group. Alleviation of symptoms was determined by data recorded in the Subject Diary. Treatment differences were assessed using a Cox Regression model with effects for current smoking behavior, treatment, and geographic region. Subjects who did not experience alleviation of symptoms were censored at the date of their last assessment. A Bonferroni adjustment for the primary comparisons of each active dose with placebo was performed.
Time Frame: Up to 14 days
Population: The intent-to-treat infected (ITTI) population included all randomized subjects who received study drug and had proven influenza by culture, PCR, or paired serology showing ≥ 4-fold increase in antibody to influenza A or B. Of the 318 subjects in the ITTI population, one subject had insufficient data to determine Time to Alleviation of Symptoms.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | Peramivir 150 mg | Peramivir 300 mg
Number analyzed (Participants) | 108 | 104 | 105
Hours | 136.2 [114.3 to 165.8] | 114.1 [95.2 to 145.5] | 117.4 [78.0 to 135.9]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 150 mg vs Peramivir 300 mg; Test type: Superiority or Other; p = 0.377, Regression, Cox; P-value is based on the treatment parameter from the Cox Regression Model including treatment, current smoking behavior, and geographic region

2. Secondary Outcome: Time to Resolution of Fever
Description: The time to resolution of fever (defined as the number of hours from initiation of study drug until temperature is less than 37.2 degrees C [99.0 degrees F] and no antipyretic medications had been taken in the previous 12 hours) was estimated using the method of Kaplan-Meier. Differences between the treatment groups were assessed using the log rank statistic controlling for current smoking behavior. Subjects who did not have resolution of fever were censored at the time of the last assessment. No adjustment for multiple comparisons was performed.
Time Frame: Up to 14 days
Population: The ITTI population included all subjects who were randomized, received study drug, and had proven influenza by any one of the following: culture, PCR, or paired serology showing ≥ 4-fold increase in antibody to influenza A or B. Subjects were analyzed according to the treatment to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | Peramivir 150 mg | Peramivir 300 mg
Number analyzed (Participants) | 108 | 104 | 104
Hours | 58.1 [43.0 to 67.7] | 43.6 [40.9 to 49.1] | 42.9 [40.2 to 46.1]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 150 mg vs Peramivir 300 mg; Test type: Superiority or Other; p = 0.007, Log Rank — P-value is based on the log-rank statistic controlling for current smoking behavior and geographic region

3. Secondary Outcome: Time to Resumption of Ability to Perform Usual Activities
Description: The time to resumption of a subject's self-assessed ability to perform his or her usual activities was estimated using the method of Kaplan-Meier. Differences between the treatment groups were assessed using the log rank statistic controlling for current smoking behavior. Subjects who were not able to resume performance of usual activities were censored at the time of the last assessment.
Time Frame: Up to 14 days
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Peramivir 150 mg | Peramivir 300 mg
Number analyzed (Participants) | 108 | 104 | 103
Days | 10.1 [9.1 to 11.4] | 9.2 [8.1 to 11.4] | 8.3 [7.3 to 10.4]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 150 mg vs Peramivir 300 mg; Test type: Superiority or Other; p = 0.537, Log Rank — P-value is based on the log-rank statistic controlling for current smoking behavior and geographic region

4. Secondary Outcome: Change From Baseline to Day 2 in Influenza Virus Titer
Description: The change in viral titers was defined as the time-weighted change from baseline in log_10 tissue culture infective dose_50 (TCID_50/mL) and was summarized for each treatment group. The differences between the treatment groups were evaluated using a Wilcoxon Rank Sum Test controlling for current smoking behavior. Specimens for virologic culture and determination of influenza virus TCID_50/mL were obtained on Day 2 (approximately 24 hours after treatment), on Day 3 (approximately 48 hours after treatment), on Day 5 (approximately 96 hours after treatment), and on Day 9 (approximately 192 hours after treatment).
Time Frame: Baseline and approximately 24 hours after treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: log10(TCID50/mL)
Arm/Group | Placebo | Peramivir 150 mg | Peramivir 300 mg
Number analyzed (Participants) | 103 | 97 | 100
log10(TCID50/mL) | -1.50 [-5.25 to 2.50] | -2.00 [-5.25 to 2.25] | -2.25 [-5.25 to 1.25]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 150 mg vs Peramivir 300 mg; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — The differences between the treatment groups were evaluated using a Wilcoxon Rank Sum Test controlling for current smoking behavior

5. Secondary Outcome: Change From Baseline to Day 3 in Influenza Virus Titer
Description: as for outcome 4
Time Frame: Baseline and approximately 48 hours after treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: log10(TCID50/mL)
Arm/Group | Placebo | Peramivir 150 mg | Peramivir 300 mg
Number analyzed (Participants) | 104 | 98 | 98
log10(TCID50/mL) | -2.75 [-5.00 to 1.00] | -3.00 [-5.25 to 1.00] | -3.25 [-6.00 to 1.25]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 150 mg vs Peramivir 300 mg; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 4, analysis 1]

6. Secondary Outcome: Change From Baseline to Day 5 in Influenza Virus Titer
Description: as for outcome 4
Time Frame: Baseline and approximately 96 hours after treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: log10(TCID50/mL)
Arm/Group | Placebo | Peramivir 150 mg | Peramivir 300 mg
Number analyzed (Participants) | 103 | 98 | 100
log10(TCID50/mL) | -3.75 [-5.50 to -0.25] | -3.38 [-6.50 to 0.00] | -3.63 [-6.50 to 0.50]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 150 mg vs Peramivir 300 mg; Test type: Superiority or Other; p = 0.409, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 4, analysis 1]

7. Secondary Outcome: Change From Baseline to Day 9 in Influenza Virus Titer
Description: as for outcome 4
Time Frame: Baseline and approximately 192 hours after treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: log10(TCID50/mL)
Arm/Group | Placebo | Peramivir 150 mg | Peramivir 300 mg
Number analyzed (Participants) | 103 | 97 | 100
log10(TCID50/mL) | -3.75 [-5.75 to -0.25] | -3.75 [-6.50 to 2.00] | -3.75 [-6.75 to -0.50]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 150 mg vs Peramivir 300 mg; Test type: Superiority or Other; p = 0.327, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Groups:
- Total: Total number of subjects who received at least 1 dose of study drug
Arm/Group | Placebo | Peramivir 150 mg | Peramivir 300 mg | Total
Serious Adverse Events (participants affected / at risk) | 1/114 | 0/113 | 1/115 | 2/342
Other Adverse Events (participants affected / at risk) | 31/114 | 27/113 | 25/115 | 83/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=114) | Peramivir 150 mg (N=113) | Peramivir 300 mg (N=115) | Total (N=342)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=114) | Peramivir 150 mg (N=113) | Peramivir 300 mg (N=115) | Total (N=342)
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 6 | 16
Nausea (Gastrointestinal disorders) | 7 | 7 | 9 | 23
Vomiting (Gastrointestinal disorders) | 5 | 4 | 2 | 11
Dizziness (Nervous system disorders) | 3 | 3 | 5 | 11
Syncope vasovagal (Nervous system disorders) | 4 | 2 | 0 | 6
Proteinuria (Renal and urinary disorders) | 7 | 10 | 5 | 22
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 3 | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 4
Insomnia (Psychiatric disorders) | 2 | 5 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No